CLINICAL TRIAL: NCT04317430
Title: Possible Role of Niclosamide in Patients With Diabetic Kidney Disease: Randomized Controlled Study
Brief Title: Niclosamide Role in Diabetic Nephropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Basma Mahrous El-Fatatry, Dr, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIC2020
Record Dates: First submitted 2020-03-18; First posted 2020-03-23 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Diabetic Nephropathies
Keywords: Diabetes - Niclosamide - Diabetic kidney disease
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Niclosamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Active Comparator): Niclosamide tablets 1 gram once daily
  Interventions: Drug: Niclosamide
- Control group (Placebo Comparator): Lactose tablets
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Niclosamide — Niclosamide tablets 1 gram once daily
  Arms: Treatment group
Drug: Placebo oral tablet — lactose tablets
  Arms: Control group

SUMMARY:
This study is randomized, controlled, parallel, prospective clinical study will be conducted on 60 patients diagnosed with type 2 diabetes mellitus at least five years ago. Patients will be recruited from Tanta University Hospital, Tanta, Egypt.

Accepted patients will be randomized into 2 groups as the following:

Control group: 30 patients will receive maximum tolerated dose of ACEI plus placebo pills for six months Treatment group: 30 patients will receive maximum tolerated dose of ACEI plus niclosamide tablets 1 gram once daily for six months The primary end point will be the change in Urinary albumin to creatinine ratio (UACR) and estimated glomerular filtration rate (eGFR) after six months of treatment

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 2 diabetes mellitus at least 5 years ago
* Stage 2 and 3 diabetic nephropathy (persistent micro- or macroalbuminuria with urinary albumin creatinine ratio (UACR) >30mg/g) despite treatment with maximum tolerated dose of ACE inhibitors for at least 8 weeks prior to the screening
* Hemoglobin A1c > 6.5 % with regular use of insulin and/or oral glucose lowering agents

Exclusion Criteria:

* Type 1 diabetes mellitus
* Severe renal impairment (eGFR< 30 mL/min/1.73 m2 at screening)
* Pregnant or lactating women
* Chronic heart failure
* Inflammatory or autoimmune disease
* History of kidney disease other than diabetic nephropathy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Change in urinary albumin creatinine ratio (UACR) | 6 months
Estimated glomerular filtration rate (eGFR) | After 6 months

SECONDARY OUTCOMES:
Change of Urinary matrix metalloproteinase-7 (MMP-7) level | 6 months
Change of Urinary podocalyxin level | 6 months

OTHER OUTCOMES:
Change of Urinary 8-hydroxy-2' -deoxyguanosine (8-OHdG) level | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Pharmacy, Tanta University, Tanta, Egypt

REFERENCES:
- [Derived] El-Fatatry BM, El-Haggar SM, Ibrahim OM, Shalaby KH. Niclosamide from an anthelmintic drug to a promising adjuvant therapy for diabetic kidney disease: randomized clinical trial. Diabetol Metab Syndr. 2023 Feb 16;15(1):22. doi: 10.1186/s13098-023-00995-1. PMID 36793092